CLINICAL TRIAL: NCT02354339
Title: Effect of Irvingia Gabonensis Administration on Metabolic Syndrome, Insulin Secretion and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-IGABONENSIS
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome; Irvingia gabonensis; African mango; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — dikanut

STUDY DESIGN:
Intervention Model Description: This is a study with two groups of patients with metabolic syndrome. One group received Irvingia Gabonensis and the other received placebo as control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irvingia gabonensis (Experimental): Irvingia gabonensis will be administered 150 mg before breakfast and 150 before dinner during 12 weeks
  Interventions: Dietary Supplement: Irvingia gabonensis
- Placebo (Placebo Comparator): Placebo will be administered 150 mg before breakfast and 150 before dinner during 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Irvingia gabonensis — Intervention will be administered 30 minutes before meals
  Other Names: African mango
  Arms: Irvingia gabonensis
Other: Placebo — Intervention will be administered 30 minutes before meals
  Other Names: calcined magnesia
  Arms: Placebo

SUMMARY:
The metabolic syndrome is a high prevalence disease worldwide. About a quarter of the adult population suffers from the disease and predispose the onset of diseases like cardiovascular disease and diabetes mellitus type 2.

The first line of treatment for metabolic syndrome is diet and exercise but patients have a low attachment to the treatment, so pharmacologic therapy is required. There is no a single drug that could help to the treatment of all metabolic syndrome components.

Irvingia gabonensis, better known as African mango, is widely consumed in central and western Africa, mainly the fruit and seeds. Besides being part of the diet of African the seeds have been used for the treatment of diseases such as dysentery, diabetes and as an analgesic.

Resent investigations have demonstrated that an extract of African mango seeds induce significantly weight loss in subjects with obesity, and also improves some biochemical parameters such as glucose and the lipid profile.

The aim of this study is to evaluate the effect of Irvingia gabonensis on metabolic syndrome, insulin secretion and insulin sensitivity.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, clinical trial is going to be carried out in 24 patients of both sexes aged between 30 and 60 years, with diagnosis of metabolic syndrome according to the modified International Diabetes Federation (IDF) criteria (without diabetes and without previous treatment for metabolic syndrome components).

The patients will be assigned randomly into two groups of 12 patients each. The patients will receive 150 mg of Irvingia gabonensis before breakfast and dinner (300 mg per day) or placebo during 12 weeks.

Waist circumference, triglycerides, high density lipoproteins (HDL-c) and blood pressure will be evaluated before and after intervention in both groups.

First phase of insulin secretion (Stumvoll index), total insulin secretion (Insulinogenic index) and Insulin sensitivity (Matsuda index) will be calculated from the concentration of glucose and insulin obtained from an Oral Glucose Tolerance Test.

Data from statistical analysis will be presented through measures of central tendency and dispersion, mean and standard deviation for quantitative variables and frequencies and percentages for qualitative variables. Qualitative variables will be analyzed by X2. The inter group differences will be analyzed through Mann-Whitney U test and Wilcoxon Test for intra-group differences. Statistical significance will be considered with a p<0.05.

This protocol was approved by a local ethics committee and written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Metabolic syndrome according IDF modified criteria
* Waist circumference: Men ≥90 cm, women ≥80 cm

And two of the following criteria:

* HDL-C: Men ≤40 mg/dL, women ≤50 mg/dL
* Fasting glucose ≥100 mg/dL
* Triglycerides ≥150 mg/dL
* Blood pressure ≥130/85 mmHg
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Known hypersensibility to Irvingia gabonensis
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid disease
* Previous treatment for the metabolic syndrome components
* Body mass index ≥ 39.9 kg/m2
* Fasting glucose ≥126 mg/dL
* Triglycerides ≥ 500 mg/dL
* Total cholesterol ≥ 240 mg/dL
* LDL-C ≥190 mg/dL
* Blood pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapéutica Experimental y Clínica, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Irvingia Gabonensis | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irvingia Gabonensis | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (7.1) | 47.8 (6.1) | 47.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] | 6.04 (0.7) | 5.9 (0.5) | 5.9 (0.6)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.5 (1.2) | 2.2 (0.6) | 2.4 (0.9)
High Density Lipoproteins (HDL-c) [Mean (Standard Deviation); unit: mmol/L] | 1.4 (0.3) | 1.6 (0.4) | 1.5 (0.4)
Systolic blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125.3 (13.0) | 128.4 (8.5) | 126.8 (10.9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.9 (7.4) | 82.7 (8.0) | 80.8 (7.8)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 94.0 (8.0) | 96.9 (9.0) | 95.5 (8.5)
First phase of insulin secretion [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 1306 (1500) | 2036 (2115) | 1670.9 (1831.0)
Total insulin secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
  index | 0.5 (0.2) | 0.8 (0.5) | 0.63 (0.37)
Total insulin sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 2.8 (1.8) | 1.9 (0.9) | 2.3 (1.5)
Body weight [Mean (Standard Deviation); unit: kilograms] | 80.6 (13.0) | 78.5 (9.2) | 79.5 (11.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (4.4) | 31.2 (3.9) | 31.6 (4.1)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.7 (0.6) | 5.4 (0.7) | 5.5 (0.7)
Low density lipoproteins (LDL-c) [Mean (Standard Deviation); unit: mmol/L] | 3.4 (1.0) | 3.0 (0.9) | 3.2 (0.7)
Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] | 27.0 (12.2) | 33.8 (27.1) | 30.4 (20.8)
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] | 27.5 (16.7) | 33.9 (20.4) | 30.7 (18.5)
Creatinine [Mean (Standard Deviation); unit: umol/L] | 70.7 (17.7) | 70.7 (17.7) | 70.7 (17.7)
Uric acid [Mean (Standard Deviation); unit: umol/L] | 374.7 (148.7) | 392.6 (59.5) | 383.7 (110.0)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose Levels at Week 12
Description: Fasting glucose will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 5.7 (0.7) | 5.9 (0.7)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of fasting glucose on Irvingia gabonensis group; Test type: Superiority; p = 0.240, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of fasting glucose on placebo group; Test type: Superiority; p = 0.850, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

2. Primary Outcome: Triglycerides Levels at Week 12
Description: Triglycerides will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 11
mmol/L | 2.0 (1.1) | 2.4 (1.8)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of triglycerides on Irvingia gabonensis group; Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of triglycerides on placebo group; Test type: Superiority; p = 0.391, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

3. Primary Outcome: High Density Lipoprotein (HDL-C) Levels at Week 12
Description: The HDL-C will be evaluated at baseline and week 12 with enzymatic-colorimetric techniques
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 1.9 (0.4) | 1.5 (0.2)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of HDL-c on Irvingia gabonensis group; Test type: Superiority; p = 0.206, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of HDL-c on placebo group; Test type: Superiority; p = 0.721, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

4. Primary Outcome: Systolic Blood Pressure at Week 12
Description: The systolic and blood pressure will be evaluated at baseline and at week 12 with a digital sphygmomanometer
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 123.5 (10.6) | 126.5 (12.1)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of systolic blood pressure on Irvingia gabonensis group; Test type: Superiority; p = 0.371, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of systolic blood pressure on placebo group; Test type: Superiority; p = 0.238, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

5. Primary Outcome: Diastolic Blood Pressure at Week 12.
Description: The diastolic and blood pressure will be evaluated at baseline and at week 12 with a digital sphygmomanometer
Time Frame: Baseline. Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 77.5 (7.3) | 81.1 (11.4)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of diastolic blood pressure on Irvingia gabonensis group; Test type: Superiority; p = 0.452, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of diastolic blood pressure on placebo group; Test type: Superiority; p = 0.801, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

6. Primary Outcome: Waist Circumference at Week 12
Description: The waist circumference will be evaluated at baseline and at week 12 with a flexible validated metric tape
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
centimeters | 91.1 (8.2) | 97.3 (8.2)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of waist circumference on Irvingia gabonensis group; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of waist circumference on placebo group; Test type: Superiority; p = 0.752, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

7. Primary Outcome: First Phase of Insulin Secretion at Week 12
Description: The first phase of insulin secretion will be calculated at baseline and week 12 with the stumvoll index from concentrations of glucose and insulin obtained of an oral glucose tolerance test.
  Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
index | 1382 (1119) | 1690 (1070)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of first phase of insulin secretion on Irvingia gabonensis group; Test type: Superiority; p = 0.791, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of first phase of insulin secretion on placebo group; Test type: Superiority; p = 0.910, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

8. Primary Outcome: Total Insulin Secretion at Week 12
Description: Total insulin secretion will be calculated at baseline and week 12 with the insulinogenic index from concentrations of glucose and insulin obtained of an oral glucose tolerance test.
  The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
index | 0.57 (0.20) | 0.8 (0.3)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of total insulin secretion on Irvingia gabonensis group; Test type: Superiority; p = 0.458, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of total insulin secretion on placebo group; Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

9. Primary Outcome: Total Insulin Sensitivity at Week 12
Description: Insulin sensitivity will be calculated at baseline and week 12 with the stumvoll index from concentrations of glucose and insulin obtained of an oral glucose tolerance test.
  Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
index | 3.5 (3.7) | 1.9 (1.2)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of insulin sensitivity on Irvingia gabonensis group; Test type: Superiority; p = 0.470, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of insulin sensitivity on placebo group; Test type: Superiority; p = 0.807, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

10. Secondary Outcome: Body Weight at Week 12
Description: The body weight will be measured at baseline and week 12 with a bioimpedance balance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
kilograms | 80.5 (12.8) | 79.0 (9.2)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of body weight on Irvingia gabonensis group; Test type: Superiority; p = 0.604, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of body weight on placebo group; Test type: Superiority; p = 0.350, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

11. Secondary Outcome: Body Mass Index at Week 12
Description: The body mass index will be calculated at baseline and week 12 with the Quetelet index
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2 | 32.0 (4.3) | 31.4 (3.8)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of BMI on Irvingia gabonensis group; Test type: Superiority; p = 0.727, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of BMI on placebo group; Test type: Superiority; p = 0.229, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

12. Secondary Outcome: Total Cholesterol at Week 12
Description: Total cholesterol will be estimated bye standardized techniques at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 5.8 (0.9) | 5.5 (0.7)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of total cholesterol on Irvingia gabonensis group; Test type: Superiority; p = 0.151, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of total cholesterol on placebo group; Test type: Superiority; p = 0.955, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

13. Secondary Outcome: Low Density Lipoproteins (LDL-C) at Week 12
Description: The LDL-C will be calculated at baseline and week 12 with the Friedewald formula
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 3.2 (0.9) | 2.8 (0.8)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of LDL-c on Irvingia gabonensis group; Test type: Superiority; p = 0.350, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of LDL-c on placebo group; Test type: Superiority; p = 0.470, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

14. Secondary Outcome: Aspartate Aminotransferase at Week 12
Description: The aspartate aminotransferase will be determinated by standardized techniques at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
U/L | 27.5 (15.8) | 27.8 (16.4)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of AST on Irvingia gabonensis group; Test type: Superiority; p = 0.910, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of AST on placebo group; Test type: Superiority; p = 0.436, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

15. Secondary Outcome: Alanine Aminotransferase at Week 12
Description: The alanine aminotransferase will be determinated by standardized techniques at baseline and week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
U/L | 27.3 (14.1) | 31.9 (23.7)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of ALT on Irvingia gabonensis group; Test type: Superiority; p = 0.989, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of ALT on placebo group; Test type: Superiority; p = 0.949, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

16. Secondary Outcome: Creatinine at Week 12
Description: Creatinine levels will be measured at baseline and week 12 with standardized techniques
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
umol/L | 61.9 (17.7) | 70.7 (17.7)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of creatinine on Irvingia gabonensis group; Test type: Superiority; p = 0.095, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of creatinine on placebo group; Test type: Superiority; p = 0.401, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

17. Secondary Outcome: Uric Acid at Week 12
Description: Uric acid levels will be measured at baseline and week 12 with standardized techniques
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Irvingia Gabonensis | Placebo
Number analyzed (Participants) | 12 | 12
umol/L | 345.0 (53.5) | 404.5 (119.0)
Statistical Analysis 1: Comparison: Irvingia Gabonensis; Results showed in this section are the result of the differences between baseline and final values of uric acid on Irvingia gabonensis group; Test type: Superiority; p = 0.910, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05
Statistical Analysis 2: Comparison: Placebo; Results showed in this section are the result of the differences between baseline and final values of uric acid on placebo group; Test type: Superiority; p = 0.791, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 12 weeks of the study.
Arm/Group | Irvingia Gabonensis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irvingia Gabonensis (N=12) | Placebo (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes